CLINICAL TRIAL: NCT01502241
Title: Temozolomid (One Week on/One Week Off) Versus Strahlentherapie in Der Primärtherapie Anaplastischer Astrozytome Und Glioblastome Bei älteren Patienten: Eine Randomisierte Phase III-Studie (Methvsalem)
Brief Title: Phase III Trial of Primary Radio- or Chemotherapy in Malignant Astrocytoma of the Elderly
Acronym: Methusalem
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Wolfgang Wick, Chairman and Director Neurooncology, Heidelberg University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NOA-08; 05-01 (Registry Identifier: German Cancer Society)
Record Dates: First submitted 2011-12-24; First posted 2011-12-30 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Glioblastoma; Anaplastic Astrocytoma
Keywords: elderly; brain tumors; MGMT; chemotherapy; Newly diagnosed; patients > 65 years
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Brain Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiotherapy (Active Comparator): 6 weeks standard partial brain treatment.
  Interventions: Radiation: Radiotherapy of the partial brain.
- Temozolomide (Experimental): Temozolomide in a one week on/one week off schedule per Wick et al. 2004 and A. Wick et al. 2007
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — 100 mg/m2 per day on seven out of fourteen days.
  Arms: Temozolomide
Radiation: Radiotherapy of the partial brain. — 60 Gy in 30 fractions à 2 Gy.
  Arms: Radiotherapy

SUMMARY:
The study aims to optimize the treatment of elderly subjects (> 65) with anaplastic astrocytoma and glioblastoma. Current treatment policies tend to be no more than palliative. There is no consensus as to how radical the surgery should be. Involved-field radiotherapy is the treatment most likely to be accepted apart from supportive and palliative measures. The role of chemotherapy is barely defined. Study data available to date does not suggest that this patient population would benefit from combined radiochemotherapy. The aim of the study is to verify the hypothesis that first-line chemotherapy with one week on/one week off temozolomide is not inferior to extended-field radiotherapy in the first-line treatment of anaplastic astrocytoma and glioblastoma in the elderly (> 65 age group). The primary endpoint is median survival, as life expectancy is limited to several months. Secondary endpoints are response rates in both arms (CR, PR, MacDonald et al. 1990), median progression-free survival, 1-year and 2-year survival rates, definition of MGMT as molecular genetic prognostic or predictive markers, and quality of life. Theoretically, it should be possible to preserve quality of life in the first-line chemotherapy arm of the study.

DETAILED DESCRIPTION:
This study is a prospective, randomized Phase III intervention study. Following histological documentation of the diagnosis by biopsy or resection of an anaplastic astrocytoma or glioblastoma, patients will be randomized either to receive postoperative extended-field radiotherapy (arm A) or to receive postoperative chemotherapy with temozolomide (arm B). Randomization will be done for all sites at the CRO, Alcedis GmbH.

For patients intending to participate in the study, the procedure is as follows:

* Request a reference neuropathological review from the brain tumor reference center in Bonn (Prof. Dr. G. Reifenberger) through the local neuropathology department. This review need not be present at randomization because anaplastic astrocytoma and glioblastoma cases are eligible
* Contact: Prof. Dr. W. Wick, Dep. Neurooncology, National Center for Tumor Diseases and Neurology Clinic, University of Heidelberg, wolfgang.wick@med.uni-heidelberg.de or CRO: Alcedis, Giessen at Alcedis GmbH, I. Helm, Winchester Str. 2, 35394 Gießen, Tel.: 0641 944360, Fax: 0641 94436 70, E-mail: ihe@alcedis.de
* Provide written confirmation that the patient signed the ethics committee-approved consent form
* Submit the registration form and a copy of the EORTC-QLQ given in Annexes

In subjects with progressive or recurrent disease, the investigating site will verify whether specific tumor treatment is justified. If yes, chemotherapy with temozolomide is recommended in arm A, possibly after further surgery. Subjects in arm B will receive radiotherapy, possible after further surgery. As all-cause mortality is the primary endpoint, all therapeutic measures following first-line therapy should be documented.

If study treatment is discontinued (first-line therapy) because of progressive disease or if progression occurs after completion of study treatment, the pertinent images should be submitted to the reference center for neuroradiology in Tübingen for reference review.

The treatment modalities employed in the study are chemotherapeutic and radiotherapeutic procedures licensed in the Federal Republic of Germany for use in human subjects. Temozolomide is currently licensed for treating subjects with recurrent disease and since 2006 in newly diagnosed glioblastoma together with radiotherapy. The time allotted for the individual treatment sections is 6 weeks for radiotherapy, while chemotherapy will be continued until progression or unacceptable adverse effects occur. The precise chemotherapy sequence is shown in the protocol. The criteria for withdrawal from the study are defined in in the protocol. Four years is the period scheduled for recruiting all patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed supratentorial anaplastic astrocytoma or glioblastoma
* Age > 65
* Karnofsky performance score > 60%
* Neutrophilic granulocyte count > 1500/µl
* Platelet count > 100 000/µl
* Hemoglobin > 10 g/dl
* Serum creatinine < 1.5 times the lab's upper normal limit
* AST or ALT < 3 times the lab's upper normal limit
* Alkaline phosphatase < 3 times the lab's upper normal limit
* No previous systemic chemotherapy
* No previous radiotherapy to the brain
* Written consent

Exclusion Criteria:

* Serious medical or neurological condition with a poor prognosis
* HIV infection
* Second cancer requiring radiotherapy or chemotherapy (contact the study coordinat if necessary)
* Hypersensitivity to temozolomide
* Conditions associated with regular vomiting that might affect oral administration of the drugs
* Psychological, familial, social or geographical circumstances with major implications for compliance with the study visit schedule
* Patient was taking part in other intervention studies within a month of starting this study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 412 (Actual)
Dates: Start 2005-01; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Overall survival | 12 months
  The primary endpoint was overall survival, measured in days from surgery to death for any reason. Patients alive at the day of the last contact were censored.

SECONDARY OUTCOMES:
Event-free survival | 12 months
  Secondary efficacy end points included EFS. EFS was defined as time from surgery to first progression for patients with progression respectively to death for patients without progression. Patients without progression or death were censored at the day of the last contact. Univariate analysis of OS and EFS used Kaplan-Meier estimates21 and a Cox proportional hazard model for evaluating Hazard Ratios (HR) with 95%-confidence intervals and median OS and EFS with 95%-confidence intervals (CI).
Best response | Within the first 8 months after surgery
  Response is assessed according MacDonald Criteria based on regular 3-monthly MRI.
Molecular prognostic or predictive biomarkers | At 12 months
  Tumor tissue, fresh or paraffine-embedded, or DNA/RNA/proteins from tissue are analyzed for the status of known molecular parameters, e.g. MGMT, for a prognostic or predictive role. Further, newly discovered molecular parameters are assessed for their potential to predict outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weller, Study Director — University of Zurich; Wolfgang Wick, Principal Investigator — Heidelberg University
Locations (23):
- Germany (22):
  - University of Heidelberg, Heidelberg, Baden-Wurttemberg
  - University of Frankfurt, Frankfurt am Main, Hesse
  - Charite Berlin, Berlin
  - University of Bochum, Bochum
  - University of Bonn, Bonn
  - University of Dresden, Dresden
  - University of Düsseldorf, Düsseldorf
  - University of Erlangen, Erlangen
  - University of Essen, Essen
  - University of Freiburg, Freiburg im Breisgau
  - University of Hamburg, Hamburg
  - University of Hannover II, Hanover
  - University of Hannover, Hanover
  - University of Homburg, Homburg
  - University of Kiel, Kiel
  - University of Leipzig, Leipzig
  - University of Mainz, Mainz
  - University of Heidelberg, Mannheim
  - University of Marburg, Marburg
  - University of Regensburg, Regensburg
  - University of Tübingen, Tübingen
  - University of Ulm, Ulm
- University of Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Wick A, Kessler T, Platten M, Meisner C, Bamberg M, Herrlinger U, Felsberg J, Weyerbrock A, Papsdorf K, Steinbach JP, Sabel M, Vesper J, Debus J, Meixensberger J, Ketter R, Hertler C, Mayer-Steinacker R, Weisang S, Bolting H, Reuss D, Reifenberger G, Sahm F, von Deimling A, Weller M, Wick W. Superiority of temozolomide over radiotherapy for elderly patients with RTK II methylation class, MGMT promoter methylated malignant astrocytoma. Neuro Oncol. 2020 Aug 17;22(8):1162-1172. doi: 10.1093/neuonc/noaa033. PMID 32064499
- [Derived] Wick W, Platten M, Meisner C, Felsberg J, Tabatabai G, Simon M, Nikkhah G, Papsdorf K, Steinbach JP, Sabel M, Combs SE, Vesper J, Braun C, Meixensberger J, Ketter R, Mayer-Steinacker R, Reifenberger G, Weller M; NOA-08 Study Group of Neuro-oncology Working Group (NOA) of German Cancer Society. Temozolomide chemotherapy alone versus radiotherapy alone for malignant astrocytoma in the elderly: the NOA-08 randomised, phase 3 trial. Lancet Oncol. 2012 Jul;13(7):707-15. doi: 10.1016/S1470-2045(12)70164-X. Epub 2012 May 10. PMID 22578793